CLINICAL TRIAL: NCT07003360
Title: Biofilm Inhibition and Remineralizing Potential of Bioactive Restorative Materials: Two-Year Randomized Clinical Trial in Class I Cavities
Brief Title: Clinical Evaluation of Bioactive Restorative Materials
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M0202025CD
Record Dates: First submitted 2025-05-12; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-02

CONDITIONS: Class I Dental Caries
Keywords: class I dental caries; bioactive materials; biofilm inhibition; remineralizing potential

STUDY DESIGN:
Who Masked: Investigator
Masking Description: * The teeth will be divided randomly into four main groups according to the restorative material will be used:
  * Each main group (n=10) depending on the material that will be used
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- application of beautiful blukfill II shofu composite (Active Comparator): Operative procedures were performed under local anesthesia and rubber dam isolation. Cavities were prepared using round diamond points (for enamel) and straight fissure and round carbide burs (for cutting in dentin) in a high-speed handpiece . Cavities were prepared following common principles for moderate to large class I adhesive resin composite restorations.
  cavities without a liner, beautiful blukfill II shofu composite were placed in bulk (a maximum 4mm thickness layer) with manual filling instruments and burnishers and cured for 40 seconds. Occlusal adjustments were performed using fine grit yellow-coded tapered with round ends and flame-shaped diamond stones (Komet, USA).
  Polishing was done using rubber points and polishing brushes (Occlubrush, Kerr, Switzerland) operated at low-speed with water coolant and minimal pressure.
  Interventions: Procedure: application of beautiful blukfill II shofu composite
- application of Ivoclar vivadent bulkfill composite (Active Comparator): Operative procedures were performed under local anesthesia and rubber dam isolation. Cavities were prepared using round diamond points (for enamel) and straight fissure and round carbide burs (for cutting in dentin) in a high-speed handpiece .Cavities were prepared following common principles for moderate to large class I adhesive resin composite restorations.
  cavities without a liner, Ivoclar vivadent bulkfill composite were placed in bulk (maximum 4mm thickness layer) with manual filling instruments and burnishers, and cured for 40 seconds ,Occlusal adjustments were performed using fine grit yellow-coded tapered with round end and flame-shaped diamond stones (Komet, USA).
  Polishing was done using rubber points and polishing brushes (Occlubrush, Kerr, Switzerland) operated at low-speed with water coolant and minimal pressure.
  Interventions: Procedure: application of Ivoclar vivadent bulkfill composite
- application of Predicta bulk fill composite (Active Comparator): Operative procedures were performed under local anesthesia and rubber dam isolation. Cavities were prepared using round diamond points (for enamel) and straight fissure and round carbide burs (for cutting in dentin) in a high-speed handpiece .Cavities were prepared following common principles for moderate to large class I adhesive resin composite restorations.
  cavities without a liner, Predicta bulk fill composite were placed in bulk (maximum 4mm thickness layer) with manual filling instruments and burnishers, and cured for 40 seconds ,Occlusal adjustments were performed using fine grit yellow-coded tapered with round end and flame-shaped diamond stones (Komet, USA).
  Polishing was done using rubber points and polishing brushes (Occlubrush, Kerr, Switzerland) operated at low-speed with water coolant and minimal pressure.
  Interventions: Procedure: application of Predicta bulk fill composite
- application of Stela self-cure bulk fill composite (Active Comparator): Operative procedures were performed under local anesthesia and rubber dam isolation. Cavities were prepared using round diamond points (for enamel) and straight fissure and round carbide burs (for cutting in dentin) in a high-speed handpiece .Cavities were prepared following common principles for moderate to large class I adhesive resin composite restorations.
  cavities without a liner, Stela self-cure bulk fill composite placed in bulk (maximum 4mm thickness layer) with manual filling instruments and burnishers, and cured for 40 seconds , Occlusal adjustments were performed using fine grit yellow-coded tapered with round end and flame-shaped diamond stones (Komet, USA).
  Polishing was done using rubber points and polishing brushes (Occlubrush, Kerr, Switzerland) operated at low-speed with water coolant and minimal pressure.
  Interventions: Procedure: application of Stela self-cure bulk fill composite

INTERVENTIONS:
Procedure: application of beautiful blukfill II shofu composite — Operative procedures were performed under local anesthesia and rubber dam isolation. Cavities were prepared using round diamond points (for enamel) and straight fissure and round carbide burs (for cutting in dentin) in a high-speed handpiece. Remaining infected carious dentin was excavated using a hand excavator. Cavities were finished using fine grit yellow-coded tapered diamond stones. 37% phosphoric acid gel was applied for 15 seconds on enamel margins, rinsed with water for 15 seconds and cavities were air-dried with Teflon protection on dentin. Self-etching universal adhesive was actively rubbed on cavity surfaces. Light curing was performed for 20 seconds. In cavities without a liner, beautiful bluk fill II composite were placed in bulk (maximum 4mm thickness layer) and cured for 40 seconds, Occlusal adjustments were performed.
  Arms: application of beautiful blukfill II shofu composite
Procedure: application of Ivoclar vivadent bulkfill composite — Operative procedures were performed under local anesthesia and rubber dam isolation. Cavities were prepared using round diamond points (for enamel) and straight fissure and round carbide burs (for cutting in dentin) in a high-speed handpiece. Remaining infected carious dentin was excavated using a hand excavator. Cavities were finished using fine grit yellow-coded tapered diamond stones. 37% phosphoric acid gel was applied for 15 seconds on enamel margins, rinsed with water for 15 seconds and cavities were air-dried with Teflon protection on dentin. Self-etching universal adhesive was actively rubbed on cavity surfaces. Light curing was performed for 20 seconds. In cavities without a liner, Ivoclar vivadent bulkfill composite were placed in bulk (maximum 4mm thickness layer) and cured for 40 seconds, Occlusal adjustments were performed.
  Arms: application of Ivoclar vivadent bulkfill composite
Procedure: application of Predicta bulk fill composite — Operative procedures were performed under local anesthesia and rubber dam isolation. Cavities were prepared using round diamond points (for enamel) and straight fissure and round carbide burs (for cutting in dentin) in a high-speed handpiece. Remaining infected carious dentin was excavated using a hand excavator. Cavities were finished using fine grit yellow-coded tapered diamond stones. 37% phosphoric acid gel was applied for 15 seconds on enamel margins, rinsed with water for 15 seconds and cavities were air-dried with Teflon protection on dentin. Self-etching universal adhesive was actively rubbed on cavity surfaces. Light curing was performed for 20 seconds. In cavities without a liner, Predicta bulk fill composite were placed in bulk (maximum 4mm thickness layer) and cured for 40 seconds, Occlusal adjustments were performed
  Arms: application of Predicta bulk fill composite
Procedure: application of Stela self-cure bulk fill composite — Operative procedures were performed under local anesthesia and rubber dam isolation. Cavities were prepared using round diamond points (for enamel) and straight fissure and round carbide burs (for cutting in dentin) in a high-speed handpiece. Remaining infected carious dentin was excavated using a hand excavator. Cavities were finished using fine grit yellow-coded tapered diamond stones. 37% phosphoric acid gel was applied for 15 seconds on enamel margins, rinsed with water for 15 seconds and cavities were air-dried with Teflon protection on dentin. Self-etching universal adhesive was actively rubbed on cavity surfaces. Light curing was performed for 20 seconds. In cavities without a liner, Stela self-cure bulk fill composite were placed in bulk (maximum 4mm thickness layer) and cured for 40 seconds, Occlusal adjustments were performed.
  Arms: application of Stela self-cure bulk fill composite

SUMMARY:
The objectives of this study are to evaluate and compare the biofilm inhibition and re-mineralizing potential at tooth restoration interface and their 2-year clinical performance in class I cavities.The patients will be selected from the Outpatient clinic at Faculty of Dentistry, Mansoura University. Patients will be informed about the steps of the study, whom will approve, will sign a written consent form. The form and protocol will be approved by the Ethics Committee. Each patient should have 4 frank carious dentinal lesions (ICDAS score 4 or 5) in posterior teeth. A periapical radiograph will be performed to evaluate the extension of the carious lesion and to ensure that there is no radiolucency in the periapical or furcation area. The teeth have to be vital, not sensitive to percussion and/or spontaneous pain. The patients will be required to have complete and normal occlusion as well as good oral hygiene.

DETAILED DESCRIPTION:
This study will be intended to evaluate and compare the biofilm inhibition and re-mineralizing potential at tooth restoration interface and their 2-year clinical performance in class I cavities.

Null hypothesis This study will be designed to test the null hypothesis that there will be no significant difference in neither biofilm inhibition nor remineralizing potential at tooth-restoration interface of the used tested materials. Also, that there will be no significant difference in the 2-year clinical outcomes of the bioactive restorative materials in class I cavities.

Sample size calculation was based on clinical performance according to FDI criteria between different bioactive restorative materials that was retrieved from previous research.19 Using G power program version 3.1.9.7 to calculate sample size, using 2-tailed test, α error =0.05 and power = 80%, the total calculated sample size will be 30 cases at least in each group Patient selection The patients will be selected from the Outpatient clinic at Faculty of Dentistry, Mansoura University. Patients will be informed about the steps of the study, whom will approve, will sign a written consent form. The form and protocol will be approved by the Ethics Committee. Each patient should have 4 frank carious dentinal lesions (ICDAS score 4 or 5) in posterior teeth. A periapical radiograph will be performed to evaluate the extension of the carious lesion and to ensure that there is no radiolucency in the periapical or furcation area. The teeth have to be vital, not sensitive to percussion and/or spontaneous pain. The patients will be required to have complete and normal occlusion as well as good oral hygiene.

Study Design:

The total number of patients will be 30 patients. Each patient will receive restorative materials studied in this investigation.

Clinical procedures All restorations will be done by a single experienced operator and with proper magnification aids. The restorative procedures will be performed under local anesthesia and rubber dam isolation. Cavity preparations for resin composite restoration will be prepared using high speed handpiece.

Evaluation procedures All restorations will be clinically evaluated immediately after finishing and polishing (baseline), 6 months, 12 months, 18 months and finally after 24 months by two independent examiners. If any restoration failed, repair or replacement of the restoration will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with four primary occlusal caries of upper or lower posterior teeth.

  * Patients must have a good oral hygiene;
  * Patients with tooth gives a positive response to testing with an electric pulp tester
  * Patients with normal and full occlusion,
  * Patients with opposing teeth should be natural with no restorations.

Exclusion Criteria:

* • High caries risk patients with extremely poor oral hygiene

  * Patients involved in orthodontic treatment or periodontal surgery,
  * Patients with periodontally involved teeth (chronic

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-02 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative hypersensitivity/pulp status | Two years after restoration
  Postoperative hypersensitivity/pulp status.The postoperative hypersensitivity/pulp status will be assessed based on the updated FDI criteria
  - Intensity was assessed with Visual Analogue Scale. Postoperative sensitivity was evaluated by blowing a stream of compressed air for 3 seconds at a distance of 2-3 cm from the restoration. -Vitality was tested with application of cold (dry ice) and compared the reaction with the adjacent vital teeth . This parameter is evaluated by scoring the pain experienced during chewing and/or with cold or warm food items, as reported by the patient. The criteria consist of five scores: scores 1-3 indicate success, score 4 indicates the need for restoration repair, and score 5 indicates the need for restoration replacement.
Marginal adaptation | Two years after restoration]
  The marginal adaptation will be evaluated through visual examination using a - A magnifying aid (loupe 4.5 x) was used for evaluation. Two special probes with different blunt tips (150 and 250 μm). This assessment will be conducted according to the updated FDI criteria. The criteria consist of five scores: scores 1- 3 indicate success, score 4 indicates the need for restoration repair, and score 5 indicates the need for restoration replacement.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Mansoura University, Egypt, Al Mansurah, Dakahliya, Egypt,, Egypt